CLINICAL TRIAL: NCT05042713
Title: The Effect of Use of Reciprocation and Rotational Single File Systems With the OneFlare Coronal Flaring Instrument on Postoperative Pain
Brief Title: The Effect of Using Different Single File Systems With Coronal Flaring Instruments on Postoperative Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Esin Özlek, Asist. Prof., Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05/22.06.2021
Record Dates: First submitted 2021-08-25; First posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Pain
Keywords: root canal; coronal flaring; single file system; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Patients will be divided into 4 groups according to the file systems to be used in root canal treatment; Group 1: Wave One Gold Group 2: One Flare + Wave One Gold Group 3: One Curve Group 4: One Flare + One Curve.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Wave One Gold (Active Comparator): The Wave One Gold file will be used with the VDW endodontic motor (VDW) in accordance with the manufacturer's recommendations.
  Interventions: Other: WaveOne Gold, One Curve, OneFlare
- One Flare and Wave One Gold file system (Active Comparator): The One Flare file will be used with a rotational speed of 300 rpm and 3 N/cm torque at a working length of 3 mm. After the Wave One Gold file will be used with the VDW endodontic motor (VDW) in accordance with the manufacturer's recommendations.
  Interventions: Other: WaveOne Gold, One Curve, OneFlare
- One Curve (Active Comparator): The One Curve file (Size 25) will be used in the VDW endodontic motor (VDW) in continuous rotation at 300 rpm and 2.5 Ncm torque in accordance with the manufacturer's recommendations.
  Interventions: Other: WaveOne Gold, One Curve, OneFlare
- One Curve with One Flare (Active Comparator): The One Flare file will be used with a rotational speed of 300 rpm and 3 N/cm torque at a working length of 3 mm. After the One Curve file (Size 25) will be used in the VDW endodontic motor (VDW) in continuous rotation at 300 rpm and 2.5 Ncm torque in accordance with the manufacturer's recommendations.
  Interventions: Other: WaveOne Gold, One Curve, OneFlare

INTERVENTIONS:
Other: WaveOne Gold, One Curve, OneFlare — During the endodontic treatment of molar teeth diagnosed with irreversible pulpitis, the effect on postoperative pain when single file systems with rotational (OneCurve) and reciprocal (WaveOne Gold) kinematics are used with and without coronal flaring instrument (OneFlare) will be compared.

SUMMARY:
Pain after root canal treatment is an important problem that affects the quality of life of patients. Common factors affecting the formation of pain after root canal treatment include insufficient root canal shaping, irrigation solution extrusion, intracanal medicament extrusion, hyperocclusion, missed canals, presence of pre-procedural pain, presence of periapical pathology, and extrusion of apical debris . It has been reported that the file systems and instrumentation technique used in root canal preparation affect apical extrusion, which is the main cause of postoperative pain . It has been reported that single-file systems introduced to the market to shorten root canal treatment time cause less postoperative pain than multi-file systems. However, there are different opinions about the effect of reciprocal and rotational file systems on postoperative pain.

It has been reported that coronal flaring during root canal shaping facilitates apical access of instruments and irrigation solution. NiTi instruments generally tend to orient tissue debris coronally, coronal shaping can create a reservoir for collecting debris accumulated in the coronal portion of the root. Therefore, increasing the coronal space for debris reduces the amount of apically removed extrusion. However, single file systems do not have a coronal flaring file and canal preparation is completed with a single file. An increased amount of apical extrusion may occur due to insufficient coronal shaping during canal preparation using single-file systems.

In this study, the effect of the use of coronal flaring file together with rotational and reciprocal single file systems on postoperative pain will be investigated, since there are different results about the effects of rotational and reciprocal file systems on postoperative pain, and although it has been reported that coronal flaring reduces apical extrusion, there is no study that determines the effect on postoperative pain. Thus, it is aimed to reduce the pain after root canal treatment and to have a more comfortable and painless process after the procedure.

DETAILED DESCRIPTION:
The study is planned to be conducted on a total of 80 patients aged between 18-45 who were diagnosed and followed up in Van Yüzüncü Yıl University, Faculty of Dentistry, Department of Endodontics. Patients with no systemic disease, diagnosis of irreversible pulpitis, single rooted and single canal lower premolar tooth will be included in the case group. Patients with resorption and calcification in the roots of their teeth, incomplete root development, pregnant and lactating patients, who have taken analgesics or anti-inflammatory drugs in the last 12 hours and cannot use a rubber dam for root canal treatment will not be included in the study. After obtaining informed consent from the patients, local anesthesia (Ultracain DS Fort, Hoechst-Marian Roussel, Frankfurt, Germany) will be administer to the tooth for which root canal treatment will be applied. Under the rubber dam isolation, the access cavity will be opened with diamond burs. Working length will be determined using a #15 K file (Mani Inc, Tochigi, Japan) and electronic apex locator (Propex Pixi, Dentsply Maillefer, Switzerland).

Patients will be divided into 4 groups according to the file systems to be used in root canal treatment;

Group 1: Wave One Gold Group 2: One Flare + Wave One Gold Group 3: One Curve Group 4: One Flare + One Curve

During the shaping process, 5.25% NaOCI and 17% EDTA will be used as irrigation solution. NaviTip irrigation needle (30-G; Ultradent Products Inc, South Jordan, USA) will be used for irrigation during shaping. After the root canal shaping is completed, the canals will be rinsed with distilled water as a final irrigation and the root canals will be filled with gutta percha and Adseal (Meta Biomed, Cheongju, North Korea) root canal sealer using the single cone technique. Teeth will be restored with composite. Patients will be prescribed 400 mg of ibuprofen anti-inflammatory medication to use in case of severe pain. The pain levels of the lines before and after the procedure will be evaluated with the VAS (Visual analogue scale) pain scale. Patients will be given a 10 cm paper ruler to record their pain levels over 6, 12, 24, 48, 72 hours and 1 week periods. Patients will be told how to score their pain levels and will be asked to mark their pain levels on the given ruler at the specified times. At the end of the 1-week period, the tables will be collected from the patients and statistical analysis will be made and interpreted for the data.

ELIGIBILITY:
Inclusion Criteria:

* Healthy persons between the ages of 18 and 45 years
* Mandibular molar teeth that were diagnosed with symptomatic irreversible pulpitis

Exclusion Criteria:

* Patients who are taken analgesic inflammatory drugs with in the last 12 hours
* Pregnancy or lactation
* Teeth with calcified canals
* Teeth with periodontal diseases
* Teeth with sensitive to percussion and palpation
* Teeth with root resorption
* Teeth with immature/open apex

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Score Scala | The change in the postoperative pain levels by the patient at the 6 hours, 12 hours, 24 hours, 48 hours, 72 hours and at the end of 1 week will be compared.
  Postoperative pain will be assessed with a visual analog score after endodontic treatment.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pedulla E, Genovesi F, Rapisarda S, La Rosa GR, Grande NM, Plotino G, Adorno CG. Effects of 6 Single-File Systems on Dentinal Crack Formation. J Endod. 2017 Mar;43(3):456-461. doi: 10.1016/j.joen.2016.10.038. Epub 2017 Jan 25. PMID 28131416